CLINICAL TRIAL: NCT05864794
Title: ValUe of Screening MRI Brain in Patients With Newly Diagnosed Stage IV Non-oncogene Addicted Non-small Cell Lung CANcer - The VULCAN Trial
Brief Title: Value of Screening MRI Brain in Stage IV Non-small Cell Lung Cancer
Acronym: VULCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NL16776
Record Dates: First submitted 2023-04-17; First posted 2023-05-18 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: brain metastasis; screening
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening population (Experimental): Patients with newly diagnosed stage IV non-oncogene addicted NSCLC, who are fit for systemic treatment and don't have any symptoms of brain disease.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI scan of the brain

SUMMARY:
Patients with newly diagnosed stage IV non-oncogene addicted NSCLC, who are fit for systemic treatment and don't have any symptoms of brain disease will undergo an MRI of the brain to screen for brain disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV metastatic NSCLC, not amenable to curative treatment.
* Fit for systemic treatment (PS 0-2) according to standard of care.
* No symptoms of brain disease disease assessed according to standard clinical care by the thoracic oncologist.

Exclusion Criteria:

* Prior/concomitant therapy for stage IV disease.
* Oncogenic diver mutation (e.g. EGFR, ALK, ROS1, RET, MET, and BRAF) with approved targeted treatment.
* Contraindications for MRI scan with contrast as per standard of care protocol of the institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical value of the MRI | up to 6 months after the MRI
  Clinical value of the MRI evaluated by the treating thoracic oncologist and assessed by questionnaires completed on three timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided